CLINICAL TRIAL: NCT03292692
Title: Empirically-Based Couple Interventions on the Web: Serving the Underserved
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of California, Los Angeles (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Brian Doss, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20120378; R01HD059802 (NIH)
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Results first posted 2018-02-12 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2018-02

CONDITIONS: Relationship, Marital; Marital Conflict

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OurRelationship (Experimental): Online Intervention
  Interventions: Behavioral: OurRelationship
- Waitlist Control (No Intervention): 2 month waiting period before couples can receive intervention

INTERVENTIONS:
Behavioral: OurRelationship — Online intervention with coach support
  Other Names: OurRelationship.com
  Arms: OurRelationship

SUMMARY:
Although several empirically-supported interventions to prevent and treat relationship distress have been developed, the majority of couples - especially high-risk couples - do not seek these face-to-face interventions. However, our pilot data indicate that large numbers of couples will seek self-administered assistance for their relationship. Additionally, unlike many in-person interventions, couples seeking self-help resources tend to have higher levels of relationship distress. Thus, to improve the reach of couple interventions, this project will translate a leading empirically-supported intervention targeting early signs of relationship distress into a Web-based format. This intervention will consist of individualized feedback and professionally-filmed video clips tailored to a couple's specific needs. By intervening effectively with a large number of couples, the resulting Web-based intervention has the potential to have a population-level impact on relationship distress, divorce, and resulting child difficulties.

In the proposed project, building off our previous pilot studies, effective translation of this in-person intervention into a Web-based format will be ensured by conducting two additional intensive pilot studies. Once final changes have been made to the website and Web-based intervention, 300 couples will be randomly assigned to a wait-list control group or an online intervention. All couples will be assessed for the initial two months; intervention couples will be assessed for one year. This project will: 1) demonstrate that couples randomly assigned to the online intervention will report higher levels of individual, child, and relationship functioning than those in the wait-list control group; 2) document the mechanisms of both active conditions; and 3) show that initial gains in those assigned to the intervention are largely maintained through one-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Currently in a heterosexual relationship
* Currently married, engaged, or cohabiting for at least 6 months
* At least one partner scoring in distressed range of relationship satisfaction (or both partners > 0.5 SD of population mean of distress).
* Living in the United States
* Both partners ages 21-64 (inclusive)

Exclusion Criteria:

* Severe Intimate Partner Violence in last 3 months
* Moderate to severe suicidal ideation in last 3 months
* Concrete plans to divorce
* Ongoing affair
* Ongoing couple therapy (or refusal to seek couple therapy for 3 months)

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2013-08-13 (Actual); Primary Completion 2014-10-18 (Actual); Study Completion 2014-10-18 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
De-identified data available to qualified researchers upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Available 2018-2020

REFERENCES:
- [Result] Doss BD, Cicila LN, Georgia EJ, Roddy MK, Nowlan KM, Benson LA, Christensen A. A randomized controlled trial of the web-based OurRelationship program: Effects on relationship and individual functioning. J Consult Clin Psychol. 2016 Apr;84(4):285-96. doi: 10.1037/ccp0000063. Epub 2016 Jan 25. PMID 26999504
- [Result] Roddy MK, Georgia EJ, Doss BD. Couples with Intimate Partner Violence Seeking Relationship Help: Associations and Implications for Self-Help and Online Interventions. Fam Process. 2018 Jun;57(2):293-307. doi: 10.1111/famp.12291. Epub 2017 Apr 20. PMID 28425562
- [Derived] Roddy MK, Stamatis CA, Rothman K, Doss BD. Mechanisms of change in a brief, online relationship intervention. J Fam Psychol. 2020 Feb;34(1):57-67. doi: 10.1037/fam0000569. Epub 2019 Aug 5. PMID 31380690
- [Derived] Doss BD, Roddy MK, Llabre MM, Georgia Salivar E, Jensen-Doss A. Improvements in coparenting conflict and child adjustment following an online program for relationship distress. J Fam Psychol. 2020 Feb;34(1):68-78. doi: 10.1037/fam0000582. Epub 2019 Aug 5. PMID 31380688

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OurRelationship | Waitlist Control
Started | 302 | 298
Completed | 264 | 260
Not Completed | 38 | 38

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OurRelationship | Waitlist Control | Total
Number analyzed (Participants) | 302 | 298 | 600
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.01 (9.54) | 36.22 (9.62) | 36.11 (9.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 149 | 300
  Male | 151 | 149 | 300
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 29 | 59
  Not Hispanic or Latino | 272 | 269 | 541
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 7
  Asian | 13 | 12 | 25
  Native Hawaiian or Other Pacific Islander | 2 | 4 | 6
  Black or African American | 62 | 57 | 119
  White | 209 | 212 | 421
  More than one race | 13 | 9 | 22
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 302 | 298 | 600

OUTCOME MEASURES:

1. Primary Outcome: Relationship Satisfaction
Description: Relationship satisfaction as measured by the total scale on the four-item version of the Couple Satisfaction Index (Funk & Rogge, 2007; doi: 10.1037/0893-3200.21.4.572). Scores on this measure range from 0-21, with higher scores indicating greater satisfaction.
Time Frame: Pre (0 weeks), Mid (3 weeks), and Post (approximately 6 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OurRelationship | Waitlist Control
Number analyzed (Participants) | 302 | 298
units on a scale
  Pre-intervention | 8.335 (3.915) | 8.37 (4.025)
  Mid-intervention | 10.63 (4.335) | 9.555 (4.53)
  Post-intervention | 12.08 (4.42) | 9.51 (4.82)
Statistical Analysis 1: Comparison: OurRelationship vs Waitlist Control; Test type: Superiority; p < 0.001, Regression, Linear; Multi-level regression; Slope = 0.372, 95% CI 2-sided [0.279 to 0.465] — Slope of intervention group compared to slope of the control group

2. Secondary Outcome: Relationship Confidence
Description: Relationship confidence as measured by 2 items from the Confidence Scale ("I believe we can handle whatever conflicts will arise in the future" and "I feel good about our prospects to make this relationship work"). Scored ranged from 0 to 12, with higher scores indicate more confidence.Cronbach's alpha = .88. These two items have been used in previous studies of couples to assess change (e.g., http://dx.doi .org/10.1177/0192513X08324388).
Time Frame: Pre (0 weeks), Mid (3 weeks), and Post (approximately 6 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OurRelationship | Waitlist Control
Number analyzed (Participants) | 302 | 298
units on a scale
  Pre-intervention | 7.94 (2.565) | 7.58 (3.185)
  Mid-intervention | 8.92 (2.495) | 8.045 (3.215)
  Post-intervention | 9.635 (2.325) | 8.05 (3.335)
Statistical Analysis 1: Comparison: OurRelationship vs Waitlist Control; Test type: Superiority; p < 0.001, Regression, Linear; Multilevel linear modeling; Slope = 0.170, 95% CI 2-sided [0.105 to 0.235] — Slope of the intervention group compared to slope of the control group

3. Secondary Outcome: Depressive Symptoms
Description: Depressive symptoms as measured by the 10-item Center for Epidemiologic Studies-Depression (CES-D) Scale (Cole, Rabin, Smith, & Kaufman, 2004). The total score was used, with possible scores ranging from 0-30. Higher scores on this measure indicate greater depressive symptoms.
Time Frame: Pre (0 weeks) and Post (approximately 6 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OurRelationship | Waitlist Control
Number analyzed (Participants) | 302 | 298
units on a scale
  Pre-intervention | 10.82 (4.24) | 10.42 (4.34)
  Post-intervention | 9.105 (3.22) | 9.895 (4.185)
Statistical Analysis 1: Comparison: OurRelationship vs Waitlist Control; Test type: Superiority; p < 0.001, Regression, Linear; Multilevel linear regression; Mean Difference (Final Values) = -2.149, 95% CI 2-sided [-2.974 to -1.324] — Multilevel linear modeling, with time modeled as change from pre-post

4. Secondary Outcome: Anxiety Symptoms
Description: Anxiety symptoms as measured by the Generalized Anxiety Disorder 7-item scale (GAD-7; Spitzer, Kroenke, Williams, & Löwe, 2006). The range of the measure is 0 to 49, with higher scores indicating greater anxiety symptoms. Cronbach's alpha in the present sample was .91.
Time Frame: Pre (0 weeks) and Post (approximately 6 weeks)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OurRelationship | Waitlist Control
Number analyzed (Participants) | 302 | 298
units on a scale
  Pre-intervention | 7.995 (5.385) | 8.24 (5.645)
  Post-intervention | 4.875 (4.5) | 6.11 (5.135)
Statistical Analysis 1: Comparison: OurRelationship vs Waitlist Control; Test type: Superiority; p = 0.002, Regression, Linear; Mean Difference (Final Values) = -1.144, 95% CI 2-sided [-1.871 to -0.417] — Multilevel linear modeling, with time modeled as change from pre to post

ADVERSE EVENTS:
Arm/Group | OurRelationship | Waitlist Control
Serious Adverse Events (participants affected / at risk) | 0/302 | 0/298
Other Adverse Events (participants affected / at risk) | 0/302 | 0/298

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No